CLINICAL TRIAL: NCT01532453
Title: Open, Multicentre, Randomised, Comparative, Prospective Trial With MD-3511356 Versus Standard Sun Protection Measures in Immunosuppressed Solid Organ Transplanted Patients for Prevention of UV-induced Carcinogenic Skin Alterations
Brief Title: Prevention of UV-induced Carcinogenic Skin Alterations in Immunosuppressed Solid Organ Transplanted Patients
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: For futility reasons and potential "loss of chance" for MD 3511356 group
Sponsor: Spirig Pharma Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SP 488/2009
Record Dates: First submitted 2012-02-09; First posted 2012-02-14 (Estimated); Results first posted 2016-01-08 (Estimated); Last update posted 2016-01-08 (Estimated); Status verified 2015-12

CONDITIONS: Actinic Keratoses; Squamous Cell Carcinomas
MeSH Terms: conditions — Keratosis, Actinic; Carcinoma, Squamous Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard Sun Protection Measures (Active Comparator): Detailed information on standardised sun protection measures and application of self-provided sunscreen products. The Investigator may decide on an individual reimbursement of patient's expenditure (out of the centre's budget).
  Interventions: Other: Standard Sun Protection Measures
- MD-3511356 (Experimental): Patients receive detailed information on standardised sun protection measures. Additionally, they will be provided free of charge with MD-3511356 for application to sun exposed skin areas once daily in the morning for 24 months. MD 3511356 lotion will be applied topically on the sun-exposed skin areas (face, neck, head, forearms and hands) in doses corresponding to the surface extent (see chapter 6.1). The dispensers will be provided with a dosage pump to allow application of reproducible amounts (each pump 0,5 g).
  Interventions: Device: MD-3511356

INTERVENTIONS:
Device: MD-3511356 — Every morning MD-3511356 should be applied liberally to those skin areas exposed to direct sunlight before exposing to the sun.
  Arms: MD-3511356
Other: Standard Sun Protection Measures — Self-provided commercially available sunscreen products, corresponding to the dosage recommendations on the product.
  Arms: Standard Sun Protection Measures

SUMMARY:
The purpose of this trial is to investigate the prevention of actinic keratoses and squamous cell carcinomas by local application of MD-3511356 in comparison to standard sun protection measures in immunosuppressed solid organ transplant recipients.

DETAILED DESCRIPTION:
This open-label multicenter, randomized, inter-individual comparative, prospective clinical trial was designed to evaluate the efficacy and safety of MD 3511356 sunscreen in preventing AK and SCC in post transplant immune-suppressed patients compared to standard of care.

The present multicenter trial is intended to contribute to the evidence that daily sun protection will have a prophylactic effect in this high risk population of chronically immune compromised patients.

ELIGIBILITY:
Inclusion Criteria:

* Out-Patients of either sex aged ≥ 40 years
* Life-expectancy of 2 years at minimum
* Solid organ-transplant recipients who received a kidney (including pancreas), liver, lung, or heart transplant
* Patients treated for 5 years with an immunosuppressant medication
* Severe sun damage of the skin
* Multiple actinic keratoses (2-5 lesions) and/or multiple dysplastic naevi
* No present squamous cell carcinoma, basal cell carcinoma or malignant melanoma; but history of cutaneous/cutaneous invasive malignancy with restitutio ad integrum is allowed
* Patients who are able to understand and provide written informed consent to participate in the clinical trial (signed informed consent) according to ICH GCP

Exclusion Criteria:

* Non-Caucasian
* Absence of sun damage i.e. no signs of AK
* Multi-organ transplantation (exception: simultaneous transplantation of kidney and pancreas)
* Evidence of systemic infection, except viral hepatitis, at the time of recruitment
* Known or supposed systemic malignant tumour or systemic chemotherapy within the last 5 years prior to randomisation
* Patients participating in a clinical trial within the last four weeks before trial
* Patients treated with the antitumour/antiangiogenetic immunosuppressant sirolimus, respectively everolimus, or acitretin or any other systemic treatment for AK at the time of randomisation
* Patients treated with a topical drug for the AK at the time of randomisation (exception: excision or Cryotherapy for hyperkeratotic lesions are allowed)
* Change of the immunosuppression-treatment less than 3 months ago or planned
* Present or planned interferon therapy (in liver transplant patients with hepatitis B/C)
* Female patients with childbearing potential with a positive pregnancy test, breast feeding, or female patients with childbearing potential without adequate contraception

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 244 (Actual)
Dates: Start 2010-11; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Claas Ulrich, MD, Principal Investigator — Klinikum der Charité Universitätsmedizin, Hauttumorzentrum Charité, D-10117 Berlin/Germany
Locations (10):
- Medizinische Universität Wien, Vienna, Austria
- Charles University Hospital, Pilsen, Czechia
- Hôpital Edouard, Lyon, France
- Germany (2):
  - Klinikum der Charité Universitätsmedizin, Berlin
  - Hautklinik am Nationalen Zentrum für Tumorerkrankungen, Heidelberg
- Beaumont Hospital, Dublin, Ireland
- Leiden University Medical Center, Leiden, Netherlands
- Universitätsspital Zürich, Dermatologische Klinik, Zurich, Switzerland
- Başkent University Faculty of Medicine, Ankara, Turkey (Türkiye)
- Queen Mary University of London, London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of 244 patients enrolled, 3 patients were considered screening failures (003-006, 005-002 and 010-027). Patient 003 006 used forbidden concomitant medication. Patient 005 002 had severe sun damage of the skin, violation of exclusion criterion #5. Patient 010 027 was re-enrolled as Patient 010 029 and later randomized to the MD-3511356 group.
Pre-assignment Details: Of 244 patients enrolled, 3 patients were considered screening failures (003-006, 005-002 and 010-027). Patient 003 006 used forbidden concomitant medication. Patient 005 002 had severe sun damage of the skin, violation of exclusion criterion #5. Patient 010 027 was re-enrolled as Patient 010 029 and later randomized to the MD-3511356 group.
Period: Overall Study
Arm/Group | Standard Sun Protection Measures | MD-3511356
Started | 81 | 160
Completed | 54 | 90
Not Completed | 27 | 70

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Sun Protection Measures | MD-3511356 | Total
Number analyzed (Participants) | 81 | 160 | 241
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.20 (9.483) | 62.29 (8.875) | 62.59 (9.075)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 45 | 61
  Male | 65 | 115 | 180

OUTCOME MEASURES:

1. Primary Outcome: Number of New Clinically Diagnosed Actinic Keratoses or Squamous Cell Carcinomas
Time Frame: 2 Years
Population: 241 patients were randomized: 160 to the MD 3511356 group and 81 to the standard care group. All 241 randomized patients received at least one dose of trial device and therefore were all included in the safety population. The Full analysis set (FAS) comprised 220 patients: 146 in the MD 3511356 group and 74 in the standard care group.
Measure: Mean (Standard Deviation); unit: new actinic keratoses or scc
Arm/Group | Standard Sun Protection Measures | MD-3511356
Number analyzed (Participants) | 74 | 146
new actinic keratoses or scc | 11.73 (14.939) | 9.88 (15.761)
Statistical Analysis 1: Comparison: Standard Sun Protection Measures vs MD-3511356; Test type: Superiority or Other; p = 0.0278, ANCOVA — Rank ANCOVA With treatment, center, gender, transplanted organ as factors and age of organ transplant as a covariable

2. Secondary Outcome: Number of Patients With New Actinic Keratoses, Squamous Cell Carcinomas or Basal Cell Carcinomas
Time Frame: 2 Years
Population: The Full analysis set (FAS) comprised 220 patients: 146 in the MD 3511356 group and 74 in the standard care group.
  For patient 10018 (MD-3511356 group) the age of first organ transplant was not computable due to missing date.
Measure: Number; unit: percentage of patients
Arm/Group | Standard Sun Protection Measures | MD-3511356
Number analyzed (Participants) | 74 | 145
percentage of patients | 83.8 | 77.2
Statistical Analysis 1: Comparison: Standard Sun Protection Measures vs MD-3511356; Test type: Superiority or Other; p < 0.05, ANCOVA; Odds Ratio (OR) = 0.579, 95% CI 2-sided [0.2703 to 1.2405]

ADVERSE EVENTS:
Arm/Group | Standard Sun Protection Measures | MD-3511356
Serious Adverse Events (participants affected / at risk) | 29/81 | 38/160
Other Adverse Events (participants affected / at risk) | 12/81 | 11/160
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Sun Protection Measures (N=81) | MD-3511356 (N=160)
squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
anemia (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1)
myocardial infarction (Cardiac disorders) | 1 (1) | 2 (2)
abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 2 (2)
diarrhea (Gastrointestinal disorders) | 1 (1) | 3 (3)
chest pain (General disorders) | 1 (1) | 2 (2)
biliary sepsis (Infections and infestations) | 2 (2) | 0 (0)
diverticulitis (Infections and infestations) | 2 (2) | 1 (1)
erysipelas (Infections and infestations) | 1 (1) | 1 (1)
gastroenteritis (Infections and infestations) | 0 (0) | 3 (3)
gastroenteritis norovirus (Infections and infestations) | 1 (1) | 1 (1)
herpes zoster (Infections and infestations) | 1 (1) | 2 (2)
influenza (Infections and infestations) | 2 (2) | 1 (1)
pneumonia (Infections and infestations) | 5 (5) | 5 (5)
respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0)
septic shock (Infections and infestations) | 1 (1) | 1 (1)
complications of transplanted kidney (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
forced expiratory volume decreased (Investigations) | 2 (2) | 1 (1)
dehydration (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
syncope (Nervous system disorders) | 1 (1) | 1 (1)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
peripheral arterial occlusive disease (Vascular disorders) | 1 (1) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Sun Protection Measures (N=81) | MD-3511356 (N=160)
pneumonia (Infections and infestations) | 5 (5) | 7 (7)
hypertension (Vascular disorders) | 7 (7) | 4 (4)

LIMITATIONS AND CAVEATS:
Trial was terminated early for futility reasons (outcome would not be changed, if trial pursued up completion) and potential "loss of chance" (which could neither be confirmed nor rejected at the time) for patients included in the MD 3511356 group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigator is granted a right to publish and present Trial Results together with other investigators of Trial and to be referred to in publications containing such results. However, investigator shall not publish or present Trial Results unless Investigator has submitted to Spirig a draft of the intended publication or presentation for review and approval.